CLINICAL TRIAL: NCT04276480
Title: Antimicrobial Therapy for Ventilator-associated Pneumonia Among Patients Colonized With Extended-spectrum Beta-lactamase-producing Enterobacteriaceae : Efficacy of a Strategy Using Piperacillin-tazobactam as Empirical Treatment.
Brief Title: Efficacy of Piperacillin-tazobactam as Empirical Antimicrobial Therapy for VAP Among ESBL-E Carriers.
Acronym: PROBATAZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2019/27
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Enterobacteriaceae Infections
Keywords: Fecal carriage; Ventilator-associated pneumonia; Piperacillin-tazobactam
MeSH Terms: conditions — Enterobacteriaceae Infections; Pneumonia, Ventilator-Associated | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The patients included will receive piperacillin-tazobactam as empirical antimicrobial therapy. The empirical microbial therapy will continue until the bacterial susceptibility profile is known.
  Interventions: Drug: Piperacillin-tazobactam

INTERVENTIONS:
Drug: Piperacillin-tazobactam — At the time of ventilator-associated pneumonia diagnosis, patients will receive an initial 4g loading dose of piperacillin-tazobactam with a continuous maintenance dose of 16g per day the first day of treatment. The dose of the piperacillin-tazobactam administered the following days will be adjusted to the renal function.
  The antimicrobial treatment will be adjusted to the narrower-spectrum agent after the antimicrobial susceptibility determination for a total length of treatment of seven days.

SUMMARY:
Antimicrobial resistance is a major threat worldwide and now concerns last-ressource antibiotics such as carbapenems. As the resistance to carbapenems is directly due to their use, their spare has become a public health emergency. Their efficacy in ventilator-associated pneumonia has never been compared to other classes of antibiotics such as piperacillin-tazobactam which can be an alternative to carbapenems.

DETAILED DESCRIPTION:
The rising antimicrobial resistance has led to more than 33,000 deaths in Europe in 2015. Among them, extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL-E) are the most frequent in Europe and carbapenems are recommended as a first line treatment by the guidelines despite the fact they are last-resource agents. Nevertheless, the overuse of carbapenems triggered the emergence of carbapenems-resistant Enterobacteriaceae (CRE). Alternatives to carbapenems are needed to treat ESBL-E infections efficiently without selecting CRE. One strategy described during the last few years is to guide the empirical antimicrobial therapy upon the fecal carriage of ESBL-E. In fact, ESBL-E fecal carriers are more often colonised in the lungs with ESBL-E and have more subsequent ESBL-E infections than non-carriers. However, the positive predictive value of ESBL-E fecal carriage for subsequent ESBL-E is only of 40% despite a negative predictive value of almost 100%. Besides, a before-after cohort study with and without ESBL-E fecal carriage screening exhibited a decrease of carbapenems consumption without any clinical harm. Several studies compared carbapenems vs alternatives after ESBL-E documentation and did not find any clinical harm either but carbapenems were almost always used before documentation. At the best of our knowledge, no study prospectively investigated an alternative to carbapenems for the empirical antimicrobial therapy (before documentation) of ventilator-associated pneumonia despite those encouraging data. This study aims to assess the relevance of piperacillin-tazobactam as the empirical antimicrobial therapy in case of a ventilator-associated pneumonia among ESBL-E fecal carriers. The treatment will be then adapted according to the susceptibility profile. The follow-up of the patients will last until 28 days after their inclusion and until their discharge from intensive care unit if it occurs later. Bacterial susceptibility to the antimicrobial treatment and clinical outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 year-old admitted to intensive care unit
* ESBL-E fecal carriage according to current screening recommendations
* Suspicion of ventilator-associated pneumonia according to ICU society guidelines

Exclusion Criteria:

* Septic shock according to Sepsis-3 classification
* Neutropenia (neutrophils count < 500/mm3)
* Known fecal carriage of Carbapenemase-producing Enterobacteriaceae or multi-drug resistant A. baumanii during the past 6 months.
* Infection with a bacteria resistant to piperacillin-tazobactam during the past 6 months
* Treatment with piperacillin-tazobactam in the 10 previous days
* Proven hypersensitivity to penicillin or tazobactam
* Pregnancy or breastfeeding
* Curatorship or guardianship
* Prisoners
* No health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Mortality in Intensive Care Unit (ICU) | at day 28 after inclusion
  Proportion of patients who died during ICU stay.

SECONDARY OUTCOMES:
Proportion of patients cured of infection on D3 and D7 after inclusion | at day 7 after inclusion
  The proportion of cured patient is defined by the combination of : hemodynamic stability, a stable or improving SOFA score AND a stable or improving Pa02 / FiO2 ratio.
Proportion of patients requiring an escalation of the probabilistic treatment of piperacillin-tazobactam to meropenem. | at day 28 after inclusion
  Therapeutic escalation of piperacillin-tazobactam to meropenem will be performed in patients in whom septic shock according to the Sepsis-3 criteria appears between inclusion and obtaining microbiological documentation and in patients in whom the condition respiratory threatens the short-term life-threatening.
Mortality at day 90 | at day 90 after inclusion
  Proportion of patients who died between D0 and D90

CONTACTS AND LOCATIONS:
Overall Officials: Laura RICHERT, Dr, Study Chair — USMR
Locations (2):
- France (2):
  - Centre hospitalier de la Côte Basque, Bayonne
  - Hopital Pellegrin, Bordeaux